CLINICAL TRIAL: NCT04464915
Title: Isopropyl Alcohol Inhalation as Anti-emetic Therapy in the Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Given the COVID-19 pandemic, there has been a temporary suspension of study activities, therefore the study has not yet been initiated.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190789-01H
Record Dates: First submitted 2020-03-06; First posted 2020-07-09 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ethanol

STUDY DESIGN:
Masking Description: The trial design is open label, given that blinding the scent of alcohol swabs is difficult. As such, no blinding of the study participants nor the research team to interventions will occur, as there will be no placebo intervention given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isopropyl alcohol swab every 10 minutes (Experimental): One deep inhalation of an isopropyl alcohol swab held 1-2cm below the nares. Intervals of administration will be every 10 minutes for a total of one hour.
  Interventions: Other: Isopropyl alcohol swab
- Isopropyl alcohol swab every 20 minutes (Experimental): One deep inhalation of an isopropyl alcohol swab held 1-2cm below the nares. Intervals of administration will be every 20 minutes for a total of one hour.
  Interventions: Other: Isopropyl alcohol swab
- No treatment arm (No Intervention): No intervention administered.

INTERVENTIONS:
Other: Isopropyl alcohol swab — Treatment will be administered by taking one deep inhalation of an isopropyl alcohol swab held 1-2cm below the nares. Intervals of administration will be every 10 minutes or every 20 minutes for a total of one hour.
  Arms: Isopropyl alcohol swab every 10 minutes; Isopropyl alcohol swab every 20 minutes

SUMMARY:
Nausea and vomiting is a common and distressing presenting complaint in Canadian emergency departments. Commonly used nausea medications have proven to be effective in certain patient populations, for example cancer patients. However, not one has been proven to be more effective that the other in the emergency department setting. In addition, many are associated with significant side effects and have the potential to interact with a patient's home medications. This limits their use in the emergency department until the patient is seen and assessed by their treating physician.

Many studies have shown that nasal inhalation of alcohol swabs is an effective therapy in relieving nausea and vomiting in post-operative patients after surgeries. The goal of this study will be to determine the effectiveness of alcohol swabs in the emergency department setting in relieving nausea and vomiting.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION:

Emerging evidence exists supporting the use of nasally inhaled isopropyl alcohol swabs as anti-emetic therapy. Multiple studies report isopropyl alcohol inhalation as an effective treatment for post-operative nausea and vomiting, with no reported adverse events. This relatively inexpensive substance is widely available in most health care settings in the form of swabs used in the routine course of delivering care as an antiseptic skin cleanser. Two previous studies in the United States have evaluated the use of inhaled isopropyl alcohol swabs in alleviating nausea and vomiting in the emergency department setting. One study in 2016 study by Beadle et. al. demonstrated superior nausea relief using inhaled isopropyl alcohol swabs compared to an inhaled placebo, while a 2018 study by April et. al. demonstrated superior nausea relief with isopropyl alcohol swabs compared with inhaled placebo and oral ondansetron.

The 2016 study by Beadle et. al. has several important limitations. This was a single center military hospital study, which only measured nausea scores 10 minutes after isopropyl alcohol swab inhalation, and lacked other important outcomes such as the number of vomiting episodes, use of rescue anti-emetics, ED length of stay and admission rates. The 2018 study by April et. al. also has limitations. Mainly, alcohol swabs were used as often as required by participants, and the dosing frequency of inhalations was not measured. They also excluded patients who had a peripheral intravenous catheter inserted on arrival, which could suggest that patients with more severe symptoms of nausea and vomiting requiring intravenous anti-emetics were excluded.

STUDY RATIONALE:

The investigator's goal is to add to the current body of evidence on the use of isopropyl alcohol in alleviating nausea and vomiting in the emergency department, particularly by determining which dosing frequency of isopropyl alcohol inhalation yields the most effective nausea relief by randomizing patients to different inhalation frequencies. This may help to guide future triage protocols enabling isopropyl alcohol inhalation before provider evaluation to improve treatment of nausea and patient satisfaction. In the current state of emergency department overcrowding, the ability to adequately control a patient's symptoms at triage may help decrease a patient's length of stay, as well as the number of patients requiring beds. In addition, from a cost-savings perspective, alcohol swabs are a relatively inexpensive therapy as compared to many commonly administered anti-emetics.

OBJECTIVES:

The objective of this study is to determine the efficacy of nasally inhaled isopropyl alcohol in alleviating nausea and/or vomiting in patients presenting to the emergency department with a chief complaint of nausea and/or vomiting. Specifically, this study will determine:

1. Nausea relief: mean reduction in nausea scores using a self-reported nausea scale comparing the pre-intervention nausea score to the final nausea score at the study endpoint.
2. Participant satisfaction: self-reported satisfaction scale measured at the study endpoint.
3. Optimal dosing frequency: compare the reduction in nausea scores among participants inhaling isopropyl alcohol swabs every 10 minutes, every 20 minutes, and to participants receiving no intervention.
4. Emergency department management: receipt of rescue anti-emetic medications and other medications (ie. analgesics, intravenous fluids).
5. Participant disposition: emergency department length of stay and admission to hospital.

OUTCOMES:

The primary outcome reflecting the efficacy of treatment is the mean nausea score reduction, using a self-reported nausea score comparing the subject's pre-intervention score to the final nausea score at the study endpoint. Nausea scores will be measured using a self-reported 10-point verbal numeric scale ranging from 1-10, labeled "no nausea" at the left end (1) and "worse nausea imaginable" at right end (10). Nausea scores will be measured at baseline before intervention, 10 minutes post-intervention, 20 minutes post-intervention, 30 minutes post-intervention, and then every 30 minutes for a total of two hours throughout the subject's emergency department visit.

The secondary outcomes reflecting the efficacy of the study intervention are participant satisfaction scores, the receipt of any rescue anti-emetic medications, emergency department length of stay, and participant disposition. Satisfaction scores will be measured using a self-reported 5-point verbal numeric scale ranging from 1-5, labeled "very unsatisfied" at the left end (1) and "very satisfied" at the right end (5).

STUDY DESIGN:

This study will be a randomized controlled trial of eligible patients presenting to the emergency department with a chief complaint of nausea and/or vomiting. Study subjects will be randomized to one of three subject arms: 1) Nasally inhaled isopropyl alcohol swabs every 10 minutes for a total of one hour; 2) Nasally inhaled isopropyl alcohol swabs every 20 minutes for a total of one hour; and 3) No intervention arm.

A convenience sample of potential study subjects will be identified by the research team during periods when available to enroll subjects. Patients will be approached while in the waiting room or shortly after arrival to their assigned emergency department room, before arrival of their treating physician and before any treatment is provided.

The allocation sequence will be generated using computer-generated random numbers using blocks of 6. Concealment will be performed using sealed, opaque envelopes.

STUDY DURATION:

Subject participation will be expected to end at the study endpoint, either after two hours of collection of nausea scores from the start of treatment or until there is administration of anti-emetics from the treating physician before the two hours is complete. There will be no further follow-up. Active study duration will be two hours for each study participant.

SAMPLE SIZE:

The minimally clinically significant difference is assumed to be 3 points on a self-reported 10-point verbal numeric scale ranging from 1-10. For α=0.25 and β=.80 using a t-test, the sample size required is 45 per participant arm (135 participants total). Imputation will be used to replace any missing data.

STATISTICAL METHODS:

All analysis will be done by the trial biostatistician. Participant baseline characteristics will be summarized with descriptive statistics with 95% confidence intervals. The primary outcome, i.e., mean reduction in nausea scores, will be analyzed using repeated measures linear regression analysis. Study arm, time and study arm by time will be included as fixed covariates and the correlation in repeated measures on the same subject over time will be modeled using a suitable covariance structure. Least square mean differences, together with 95% Confidence Intervals, will be used to express the treatment effect, comparing each of the intervention arms to the control arm. Statistical significance of each pairwise comparison will be judged at the 2.5% level to maintain the overall level at 5%. A similar approach will be used for ED lengths of stay (with transformation to improve normality if necessary). Number of vomiting episodes and receipt of antiemetic drugs will be analyzed using Poisson or logistic regression as appropriate. All analyses will be intention to treat. There will be no interim analysis completed. Imputation will be used to replace any missing data.

QUALITY CONTROL:

The study will have a quality control monitoring process and study monitor plan in place to verify that all data are accurate and complete. An internal DSMB, free of competing interests, will monitor the study and will generate a site monitoring report to detail significant findings, deviations, deficiencies, plausibility, record completeness and any corrective actions to be taken. The investigator will permit trial-related monitoring, audits, REB review, and regulatory inspection(s) by providing direct access to source data/documents.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years) presenting to the emergency department with a chief complaint of nausea and/or vomiting with a level of 3 or greater on a verbal numeric response scale (1-10).

Exclusion Criteria:

* Not able to breathe through nares (ie. rhinitis)
* Known pregnancy
* Have already received an anti-emetic within the past 24 hours (including while in emergency department triage)
* Chronic nausea (> 1 month)
* Known allergy to isopropyl alcohol
* Nasally sensitive to inhaled chemical products
* Altered mental status or underlying cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Change in nausea scores from pre-intervention to post-intervention | From the time of randomization over two hours
  Self-reported 10-point verbal numeric scale ranging from 1-10, labeled "no nausea" at the left end (1) and "worse nausea imaginable" at right end (10).

SECONDARY OUTCOMES:
Subject satisfaction score | From the time of randomization over two hours
  Self-reported 5-point verbal numeric scale ranging from 1-5, labeled "very unsatisfied" at the left end (1) and "very satisfied" at the right end (5).
Receipt of rescue anti-emetics | From the time of randomization until the time of documented emergency department disposition (either admission to hospital or discharge home
  The receipt of any rescue anti-emetics by the treating physician will be recorded, including the medication type(s), and number of doses.
Emergency department length of stay | From the time of emergency department arrival until documented emergency department disposition (either admission to hospital or discharge home)
  The subject's total emergency department length of stay (in minutes).
Subject disposition | From the time of emergency department arrival until documented emergency department disposition (either admission to hospital or discharge home
  Subject disposition from the emergency department, either admission to hospital or discharge home.

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Thiruganasambandomoorthy, MD, Principal Investigator — Senior Scientist, Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hines S, Steels E, Chang A, Gibbons K. Aromatherapy for treatment of postoperative nausea and vomiting. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD007598. doi: 10.1002/14651858.CD007598.pub2. PMID 22513952
- [Background] Beadle KL, Helbling AR, Love SL, April MD, Hunter CJ. Isopropyl Alcohol Nasal Inhalation for Nausea in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2016 Jul;68(1):1-9.e1. doi: 10.1016/j.annemergmed.2015.09.031. Epub 2015 Dec 8. PMID 26679977
- [Background] April MD, Oliver JJ, Davis WT, Ong D, Simon EM, Ng PC, Hunter CJ. Aromatherapy Versus Oral Ondansetron for Antiemetic Therapy Among Adult Emergency Department Patients: A Randomized Controlled Trial. Ann Emerg Med. 2018 Aug;72(2):184-193. doi: 10.1016/j.annemergmed.2018.01.016. Epub 2018 Feb 17. PMID 29463461
- [Background] Hesketh PJ, Kris MG, Basch E, Bohlke K, Barbour SY, Clark-Snow RA, Danso MA, Dennis K, Dupuis LL, Dusetzina SB, Eng C, Feyer PC, Jordan K, Noonan K, Sparacio D, Somerfield MR, Lyman GH. Antiemetics: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2017 Oct 1;35(28):3240-3261. doi: 10.1200/JCO.2017.74.4789. Epub 2017 Jul 31. PMID 28759346
- [Background] Furyk JS, Meek RA, Egerton-Warburton D. Drugs for the treatment of nausea and vomiting in adults in the emergency department setting. Cochrane Database Syst Rev. 2015 Sep 28;2015(9):CD010106. doi: 10.1002/14651858.CD010106.pub2. PMID 26411330
- [Background] Patanwala AE, Amini R, Hays DP, Rosen P. Antiemetic therapy for nausea and vomiting in the emergency department. J Emerg Med. 2010 Sep;39(3):330-6. doi: 10.1016/j.jemermed.2009.08.060. Epub 2009 Dec 21. PMID 20022195